CLINICAL TRIAL: NCT05406271
Title: Influence of Use of Intraoperative Fluoroscopy on the Hip Prosthesis Components Position
Brief Title: Hip Prosthesis Components Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mateusz Szymczak (Other)
Responsible Party: Sponsor-Investigator, Mateusz Szymczak, MD Phd, Independent Public Healthcare Center in Rypin
Organization: Independent Public Healthcare Center in Rypin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Hip Arthrosis
Keywords: hip prosthesis; center of rotation; offset
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Prosthesis with intraoperative fluoroscopy (Experimental)
  Interventions: Diagnostic Test: Intraoperative fluoroscopy
- Hip Prosthesis without intraoperative fluoroscopy (No Intervention)

INTERVENTIONS:
Diagnostic Test: Intraoperative fluoroscopy — Impantation of hip prosthesis with intraoperative fluoroscopy
  Arms: Hip Prosthesis with intraoperative fluoroscopy

SUMMARY:
The purpose of the study is

ELIGIBILITY:
Inclusion Criteria:

* indication for hip replacement surgery

Exclusion Criteria:

* pregnancy
* abnormal anatomy (hip dysplasia, fracture)
* previous srgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Prosthesis cup position | Day 1 after surgery
  inclination, anteversion, centre of rotation of the prosthesis cup. Measurement will be made on post x-rays

SECONDARY OUTCOMES:
Prosthesis steam position | Day 1 after surgery
  Leg length, total offset of the hip prosthesis. Measurement will be made on post x-rays

CONTACTS AND LOCATIONS:
Locations (1):
- District Hospital, Rypin, Kuyavian-Pomeranian Voivodeship, Poland